CLINICAL TRIAL: NCT01992848
Title: A Case-control Study of MicroRNAs a Potential Biomarkers for Coronary Artery Calcification (CAC) - An Additional Substudy to Determine the Relationship Between CAC and Bone Mineral Density and Markers of Bone Metabolism
Brief Title: MAP-Calcification: MicroRNAs as Potential Biomarkers for Coronary Artery Calcification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: MAP-Calcification
Record Dates: First submitted 2013-10-23; First posted 2013-11-25 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Coronary Artery Calcification; Coronary Artery Disease; Osteoporosis; Osteopenia
MeSH Terms: conditions — Coronary Artery Disease; Osteoporosis; Bone Diseases, Metabolic | interventions — Blood Specimen Collection; Diet Records

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All participants (Experimental): Venous blood sampling 4-day food diary
  1 week UV Dosimeter Peripheral Quantitative Computed Tomography of the radius
  Interventions: Other: Venous blood sampling; Other: 4-day food diary; Other: 1 week UV dosimeter; Radiation: Peripheral Quantitative Computed Tomography of the radius

INTERVENTIONS:
Other: Venous blood sampling — 40ml venous blood sampling will be undertaken during participants' attendance for CT coronary angiography (the latter being performed as part of routine clinical investigation).
Other: 4-day food diary
Other: 1 week UV dosimeter — To be worn on outerwear for one week week prior to attendance for pQCT
Radiation: Peripheral Quantitative Computed Tomography of the radius — To be performed within one month of attendance for CT coronary angiography

SUMMARY:
Coronary artery disease (CAD) remains the leading cause of mortality in the UK with an estimated 80,000 fatalities in 2010. Coronary artery calcification (CAC) is associated with atherosclerotic plaque burden and cardiovascular mortality. Mechanisms underlying isolated CAC have not been as yet been fully explained. MicroRNAs (miRNAs), known to act as regulators of gene expression, have also emerged as powerful biomarkers in the diagnosis and prognosis of cardiovascular disorders and may be used in the detection of CAC. We aim to investigate the potential for a "microRNA-signature" in patients with CAC by performing a prospective, case-controlled study to identify pathways associated with CAC in humans. Previous research has demonstrated an inverse relationship between CAC and bone mineral density (BMD), suggesting that these processes may be linked. In a further substudy we plan to define the relationship between CAC and BMD as well as a number of markers of bone metabolism.

DETAILED DESCRIPTION:
Patients will be prospectively enrolled whilst attending for elective coronary CT (computed tomography) angiography including a coronary calcium score, at the Royal Surrey County Hospital. Data regarding demographic and clinical characteristics of patients will be collected. Peripheral venous blood sampling will take place on this occasion. Coronary artery calcification scores will be estimated by a Radiologist using default software. Patients eligible for the bone metabolism substudy will be required to attend the University of Surrey for peripheral Quantitative Computed Tomography (pQCT) of bone mineral composition of the radius. In the intervening period we will ask them to complete a 4-day food diary and wear a UV dosimeter, the latter to assess typical UV exposure, for one week.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient is able to provide written, informed consent

Exclusion Criteria:

* Age > 65 years
* Diabetes mellitus
* Glomerular filtration rate ≤ 60 ml/min
* Abnormal serum calcium
* History or clinical features of cardiac failure
* Systemic inflammatory disease
* Peripheral vascular disease
* Previous history of percutaneous coronary intervention (PCI)
* Previous history of coronary artery bypass grafting (CABG)
* Previous history of reno-vascular disease
* Active infection
* Active malignancy

Additional clinical exclusion criteria for our sub-study are:

* Regular use of sunbeds
* A sun holiday one month prior to or plans for sun holiday within the study
* Use of vitamin D supplements
* Consumption of alcohol above recommended levels
* Pregnancy or planned pregnancy
* Use of a veil

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
A miRNA signature in the presence and absence of coronary artery calcification (CAC) | 12 months

SECONDARY OUTCOMES:
mRNA(messenger RNA) targets of identified miRNAs in the presence and absence of CAC | 12 months
Bone Mineral Density (BMD) in the presence and absence of CAC | 12 months
Markers of bone metabolism in the presence and absence of CAC to include: serum 25-hydroxy vitamin D, 1,25-dihydroxy vitamin D, serum calcium, albumin, parathyroid hormone, C-terminal telopeptide/CTX, and lipid profile. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mahmoudi, MBChB PhD, Principal Investigator — The University of Surrey; Chris Fry, BSc PhD, Study Director — The University of Surrey
Locations (2):
- United Kingdom (2):
  - The University of Surrey, Guildford, Surrey
  - The Royal Surrey County Hospital, Guildford, Surrey

REFERENCES:
- [Derived] Howlett P, Cleal JK, Wu H, Shah N, Horton A, Curzen N, Mahmoudi M. MicroRNA 8059 as a marker for the presence and extent of coronary artery calcification. Open Heart. 2018 Jan 31;5(1):e000678. doi: 10.1136/openhrt-2017-000678. eCollection 2018. PMID 29531756